CLINICAL TRIAL: NCT04749537
Title: The Relationship Between The Decreasing Activity, Depression And Quality Of Life In Work Productivity And Social Activities In Ankylosing Spondylitis Patients: A Randomized Controlled Trial
Brief Title: Work Productivity and Social Activities In Patients With Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IstPRMTRH-ASWP
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Ankylosing Spondylitis; Work Productivity
Keywords: Spondylitis; Ankylosing; Quality of Life; Employment
MeSH Terms: conditions — Spondylitis, Ankylosing; Spondylitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ankylosing Spondylitis: 100 patients who were diagnosed with AS between the ages of 18-65
- Healthy Volunteers: 100 healthy volunteers compatible with age.

SUMMARY:
The aim of this study is to evaluate the relationship between decrease in work productivity and social activities in patients with Ankylosing Spondylitis (AS) with disease activity, depression and quality of life together with demographic data.

DETAILED DESCRIPTION:
For this study, which is planned as a cross-sectional clinical study, 100 patients who were diagnosed with AS between the ages of 18-65 and who applied to the Istanbul Physical Therapy Rehabilitation SUAM Physical Medicine and Rehabilitation Outpatient Clinic between April 15, 2019, and April 15, 2020, and 100 healthy volunteers compatible with age. was included. Demographic data of the participants were recorded. Work productivity and activity reduction questionnaire: general health (WPAI: GH), social role participation questionnaire short form (SRPQ), short form-36 (SF-36), hospital anxiety, and depression scale (HADS), will be evaluated. Besides, if the patient group exists, laboratory results (CRP, erythrocyte sedimentation rate, HLA-B27), and bath ankylosing spondylitis functional index (BASFI), bath ankylosing spondylitis disease activity index (BASDAI), Bath ankylosing spondylitis metrology index (BASMI), visual analog scale (VAS) resting, night and activity values were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AS diagnosis between the ages of 18-65
* Healthy volunteer individuals between the ages of 18-65 without known musculoskeletal disease

Exclusion Criteria:

* Those with serious systemic diseases that may interfere with working (respiratory system, cardiovascular system, renal and metabolic diseases)
* Those with orthopedic and psychiatric diseases
* Those with inflammatory diseases other than known AS
* Pregnant
* People with disability due to the history of trauma
* Those with injury after the operation
* Those with diseases that cause neurological sequelae

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, which is planned as a cross-sectional clinical study, 100 patients who were diagnosed with AS between the ages of 18-65 and who applied to the Istanbul Physical Therapy Rehabilitation SUAM Physical Medicine and Rehabilitation Outpatient Clinic between April 15, 2019, and April 15, 2020, and 100 healthy volunteers compatible with age was included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH) | One day
  WPAI: GH measures health impact and symptom severity impact on work productivity and leave time effectiveness
Social Role Participation Questionnaire (SRPQ) | One day
  It is used to evaluate integration into society and activities in social life. It evaluates the level of participation in six social roles in two dimensions: the "experienced physical difficulties scale" and the "role performance satisfaction scale". Participants complete their satisfaction and challenges during their social roles

SECONDARY OUTCOMES:
Short Form Health Survey 36 (SF-36) | One day
  used to evaluate the quality of life
Hospital Anxiety and Depression Scale (HADS) | One day
  used to determine the risk in terms of anxiety and depression in a patient with a physical illness, and to measure the level and change of severity.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | One day
  the assessment of disease activity in patients with ankylosing spondylitis
Bath Ankylosing Spondylitis Functional Index (BASFI) | One day
  the assessment of functional status in patients with ankylosing spondylitis
Bath Ankylosing Spondylitis Metrology Index (BASMI) | One day
  the assessment of the level of spinal mobility in patients with ankylosing spondylitis
Ankylosing Spondylitis Quality of Life (ASQoL) | One day
  used to evaluate the quality of life in patients with ankylosing spondylitis
Visual Analogue Scale (VAS) | One day
  used to evaluate the pain

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Faruk Bucak, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Derya Bugdayci, Assoc Prof, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Macfarlane GJ, Shim J, Jones GT, Walker-Bone K, Pathan E, Dean LE. Identifying Persons with Axial Spondyloarthritis At Risk of Poor Work Outcome: Results from the British Society for Rheumatology Biologics Register. J Rheumatol. 2019 Feb;46(2):145-152. doi: 10.3899/jrheum.180477. Epub 2018 Nov 1. PMID 30385702
- [Background] Goh Y, Kwan YH, Leung YY, Fong W, Cheung PP. A cross-sectional study on factors associated with poor work outcomes in patients with axial spondyloarthritis in Singapore. Int J Rheum Dis. 2019 Nov;22(11):2001-2008. doi: 10.1111/1756-185X.13696. Epub 2019 Oct 1. PMID 31576680
- [Background] Sag S, Nas K, Sag MS, Tekeoglu I, Kamanli A. Relationship of work disability between the disease activity, depression and quality of life in patients with ankylosing spondylitis. J Back Musculoskelet Rehabil. 2018;31(3):499-505. doi: 10.3233/BMR-169657. PMID 29504521
- [Background] van Lunteren M, Ez-Zaitouni Z, Fongen C, Landewe R, Ramonda R, van der Heijde D, van Gaalen FA. Disease activity decrease is associated with improvement in work productivity over 1 year in early axial spondyloarthritis (SPondyloArthritis Caught Early cohort). Rheumatology (Oxford). 2017 Dec 1;56(12):2222-2228. doi: 10.1093/rheumatology/kex365. PMID 29155961
- [Background] Oude Voshaar M, van Onna M, van Genderen S, van de Laar M, van der Heijde D, Heuft L, Spoorenberg A, Luime J, Gignac M, Boonen A. Development and Validation of a Short Form of the Social Role Participation Questionnaire in Patients with Ankylosing Spondylitis. J Rheumatol. 2016 Jul;43(7):1386-92. doi: 10.3899/jrheum.151013. Epub 2016 May 15. PMID 27182067
- [Background] van Genderen S, Plasqui G, Landewe R, Lacaille D, Arends S, van Gaalen F, van der Heijde D, Heuft L, Luime J, Spoorenberg A, Gignac M, Boonen A. Social Role Participation in Patients With Ankylosing Spondylitis: A Cross-Sectional Comparison With Population Controls. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1899-1905. doi: 10.1002/acr.22907. Epub 2016 Oct 28. PMID 27059161
- [Background] Cakar E, Taskaynatan MA, Dincer U, Kiralp MZ, Durmus O, Ozgul A. Work disability in ankylosing spondylitis: differences among working and work-disabled patients. Clin Rheumatol. 2009 Nov;28(11):1309-14. doi: 10.1007/s10067-009-1249-1. Epub 2009 Aug 16. PMID 19685294
- [Background] Maksymowych WP, Gooch KL, Wong RL, Kupper H, van der Heijde D. Impact of age, sex, physical function, health-related quality of life, and treatment with adalimumab on work status and work productivity of patients with ankylosing spondylitis. J Rheumatol. 2010 Feb;37(2):385-92. doi: 10.3899/jrheum.090242. Epub 2009 Dec 1. PMID 19955052
- [Background] Deodhar AA, Dougados M, Baeten DL, Cheng-Chung Wei J, Geusens P, Readie A, Richards HB, Martin R, Porter B. Effect of Secukinumab on Patient-Reported Outcomes in Patients With Active Ankylosing Spondylitis: A Phase III Randomized Trial (MEASURE 1). Arthritis Rheumatol. 2016 Dec;68(12):2901-2910. doi: 10.1002/art.39805. PMID 27390130